CLINICAL TRIAL: NCT00667836
Title: Multi-center Project: Spinal Abnormalities in Neurofibromatosis Type1 (NF1) Patients
Status: Completed | Type: Observational
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Jacques D'Astous, Principal Investigator, Shriners Hospitals for Children
Other Study IDs: IRB_00023261
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Neurofibromatosis Type 1
Keywords: Neurofibromatosis Type 1; NF1; Spinal Anomalies
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We propose to establish a multi-center study to investigate the outcome of scoliosis and spinal abnormalities in patients with NF1.

The three specific aims of this study are:

Specific Aim 1 - To assess health status and health-related quality of life (HRQL) in children and adolescents with NF1 and scoliosis. We hypothesize that children and adolescents with NF1 and scoliosis will experience an additional burden of morbidity due to scoliosis and a downward trajectory of health status and HRQL over time.

Specific Aim 2 - To assess the natural history and short-term response to therapy in a cohort of children with NF1 and scoliosis prospectively diagnosed during the course of the four-year study period. We hypothesize that some NF1 patients with idiopathic scoliosis will modulate to the dystrophic form. We also hypothesize that NF1 patients with earlier presentation are more likely to have or modulate to the dystrophic form.

Specific Aim 3 - To assess biochemical markers of bone metabolism in NF1 individuals. We hypothesize that NF1 individuals will have statistically significant differences in biochemical markers of bone metabolism compared to controls. We also hypothesize that NF1 individuals with scoliosis will have differences in biochemical markers of bone metabolism compared to NF1 individuals without scoliosis.

DETAILED DESCRIPTION:
The three specific aims of this study are:

Specific Aim 1 - To assess health status and health-related quality of life (HRQL) in children and adolescents with NF1 and scoliosis. We hypothesize that children and adolescents with NF1 and scoliosis will experience an additional burden of morbidity due to scoliosis and a downward trajectory of health status and HRQL over time.

Specific Aim 2 - To assess the natural history and short-term response to therapy in a cohort of children with NF1 and scoliosis prospectively diagnosed during the course of the four-year study period. We hypothesize that some NF1 patients with idiopathic scoliosis will modulate to the dystrophic form. We also hypothesize that NF1 patients with earlier presentation are more likely to have or modulate to the dystrophic form.

Specific Aim 3 - To assess biochemical markers of bone metabolism in NF1 individuals. We hypothesize that NF1 individuals will have statistically significant differences in biochemical markers of bone metabolism compared to controls. We also hypothesize that NF1 individuals with scoliosis will have differences in biochemical markers of bone metabolism compared to NF1 individuals without scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* Meet NIH diagnostic criteria for NF1
* Radiographic documentation of scoliosis will be necessary for inclusion as a "scoliosis case"
* Age between 3 and 18 years

Exclusion Criteria:

* Do not have NF1

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All NF1 patients
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques D'Astous, M.D., Principal Investigator — Shriners Hospitals for Children
Locations (1):
- Shriners Hospitals for Children, Salt Lake City, Salt Lake City, Utah, United States